CLINICAL TRIAL: NCT06160713
Title: A Randomized Controlled Trial to Compare Oral Itraconazole and Standard Care Versus Standard Care Alone in Patients With Non-cystic Fibrosis Related Bronchiectasis With Chronic Aspergillus Infection in Reducing Bronchiectasis Exacerbations
Brief Title: Compare Oral Itraconazole and Standard Care Versus Standard Care Alone in Patients With Non-cystic Fibrosis Related Bronchiectasis With Chronic Aspergillus Infection in Reducing Bronchiectasis Exacerbations
Acronym: BAIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study 1291
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Bronchiectasis; Bronchiectasis Adult
MeSH Terms: conditions — Bronchiectasis | interventions — Itraconazole; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Standard care of bronchiectasis
  Interventions: Other: Standard care
- Itraconazole arm (Experimental): Supra-bioavailable- Itraconazole capsule 65 mg
  Interventions: Drug: Itraconazole 65 MG; Other: Standard care

INTERVENTIONS:
Drug: Itraconazole 65 MG — Two capsules of suba-itraconazole 65 mg twice daily for 6 months
  Arms: Itraconazole arm
Other: Standard care — Standard care for bronchiectasis

SUMMARY:
There is an intricate link between bronchiectasis and fungi. Patients with cystic fibrosis frequently manifest fungal sensitization and fungal colonization with Aspergillus fumigatus.6 Aspergillus species also has a cause-and-effect relationship with non-CF (cystic fibrosis) bronchiectasis.7, 8 In allergic bronchopulmonary aspergillosis (ABPA), Aspergillus is the cause of bronchiectasis. In contrast, in other causes of bronchiectasis, A fumigatus can theoretically promote allergic response, which may result in poor lung function, increase the risk of exacerbations, and even cause ABPA over time.9, 10 In a recent study, we found an overall prevalence of Aspergillus sensitization of 29.5% and the prevalence of chronic aspergillus infection was 76%.11 The prevalence of chronic aspergillus colonization in non-(tuberculosis) TB-non-CF fibrosis was 47.5% (49/103).11 By mechanism similar to chronic bacterial colonization, chronic aspergillus infection or aspergillus sensitization can increase the risk of bronchiectasis exacerbation. Therefore, eradication of A. fumigatus from the airways of patients with bronchiectasis would decrease the future risk of a bronchiectasis exacerbation. Notably, in ABPA, use of itraconazole and voriconazole reduce the exacerbations by reducing the fungal burden in the airways.12, 13 In this randomized trial, we will investigate whether treatment with oral itraconazole for six months would reduce the future risk of bronchiectasis exacerbation in patients with non-CF-non-ABPA bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic lung disease due to irreversible and abnormal dilatation of the bronchi. Bronchiectasis manifest with chronic cough, expectoration, hemoptysis, dyspnea, and others. Bronchiectasis can be broadly classified as genetic (cystic fibrosis [CF], ciliary dyskinesia and others) or acquired (post-infective, tuberculosis (TB), allergic bronchopulmonary aspergillosis [ABPA] and others).1 The natural course of bronchiectasis is associated with recurrent exacerbations that cause further damage and disease progression.2 Most exacerbations are caused by viral or bacterial infections, inflammation and external environment factors. Chronic bacterial infections increase the risk of bronchiectasis exacerbation.2 In a multicentric European study chronic infection with Pseudomonas aeruginosa was associated with an increased risk of exacerbation.3 Notably, change in the interaction between the bacterial microbiome by external inciting events (viral infection or air pollution) increases exacerbation risk.4 Similarly, viral infections by increasing the systemic and airway inflammation induce a bronchiectasis exacerbation.5 Airway inflammation both neutrophilic and eosinophilic are also important causes of bronchiectasis exacerbations.2 Most previous studies in non-CF bronchiectasis have not investigated the role of fungal sensitization or chronic fungal infection in causing bronchiectasis exacerbation.

There is an intricate link between bronchiectasis and fungi. Patients with cystic fibrosis frequently manifest fungal sensitization and fungal colonization with Aspergillus fumigatus.6 Aspergillus species also has a cause-and-effect relationship with non-CF bronchiectasis.7, 8 In ABPA, Aspergillus is the cause of bronchiectasis. In contrast, in other causes of bronchiectasis, A fumigatus can theoretically promote allergic response, which may result in poor lung function, increase the risk of exacerbations, and even cause ABPA over time.9, 10 In a recent study, we found an overall prevalence of Aspergillus sensitization of 29.5% and the prevalence of chronic aspergillus infection was 76%.11 The prevalence of chronic aspergillus colonization in non-TB-non-CF fibrosis was 47.5% (49/103).11 By mechanism similar to chronic bacterial colonization, chronic aspergillus infection or aspergillus sensitization can increase the risk of bronchiectasis exacerbation. Therefore, eradication of A. fumigatus from the airways of patients with bronchiectasis would decrease the future risk of a bronchiectasis exacerbation. Notably, in ABPA, use of itraconazole and voriconazole reduce the exacerbations by reducing the fungal burden in the airways.12, 13 In this randomized trial, we will investigate whether treatment with oral itraconazole for six months would reduce the future risk of bronchiectasis exacerbation in patients with non-CF-non-ABPA bronchiectasis.

Study question: Does oral itraconazole for six months reduce the bronchiectasis exacerbation in patients with non-cystic fibrosis bronchiectasis?

ELIGIBILITY:
Inclusion Criteria: adults subjects (≥13 years) with non-cystic fibrosis bronchiectasis fulfilling all the following criteria: • bronchiectasis on thin-section computed tomography (CT)

* chronic aspergillus infection defined by the presence of A.fumigatus-specific IgG ≥40 mgA/L
* clinically stable for at least three months prior to study inclusion

Exclusion Criteria:

We will exclude subjects with any of the following:

* allergic bronchopulmonary aspergillosis as the cause of underlying bronchiectasis
* cystic fibrosis
* post-tuberculosis bronchiectasis
* severe asthma
* current smokers
* active bacterial, mycobacterial (atypical or typical), or fungal (aspergillosis or mucormycosis) infections
* use of systemic antifungal drugs in past 3 months
* previous documented intolerance to itraconazole
* pregnancy
* failure to provide informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
frequency of bronchiectasis exacerbations during the study period | (12 months [6 months each of intervention and observation])
  An exacerbation will be defined as clinical deterioration for at least 48 hours and the presence of three or more of the following six features: (1) increase in cough; (2) sputum volume/consistency; (3) sputum purulence; (4) breathlessness or exercise intolerance; (5) fatigue, malaise, or fever; (6) hemoptysis; and change of bronchiectasis treatment by a physician

SECONDARY OUTCOMES:
time to first exacerbation | 12 months
  Time taken for the first exacerbation
change in the spirometric lung function (FVC) | 12 months
  Spirometry will be done to measure FVC
change in the spirometric lung function ( FEV1) | 12 months
  Spirometry will be done to measure FEV1
Change in 6 minute walk distance | 6 months
  6 minute walk test will be done at baseline and at treatment completion
Adverse events | 6 months
  Adverse events during therapy will be assessed
change in the quality of life assessed by bronchiectasis health questionnaire | 6 months
  We will use BHQ at baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chest clinic, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
It will be shared after a reasonable request to the corresponding author and obtaining proper ethics approval